CLINICAL TRIAL: NCT03032211
Title: A Feasibility Clinical Study of Osmotic Pump Treatment in Fluid Management to Achieve Optimal Fluid Balance in NYHA Class III and Ambulatory NYHA Class IV Heart Failure Patients Who Have an Estimated Glomerular Filtration Rate of > 15 to < 60 mL/Min/1.73m2
Brief Title: Optimal Balance Alfapump® System Feasibility Study
Acronym: OPTIMALBALANCE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in company strategy
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-CHF-003
Record Dates: First submitted 2016-08-11; First posted 2017-01-26 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2018-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: • Prospective, non-randomized, open label, single-arm study to evaluate the safety and feasibility of the use of the alfapump® system in New York Heart Association (NYHA) Class III and ambulatory NYHA Class IV heart failure patients with a history of at least one hospitalization for fluid management within the previous year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Alfapump
  Interventions: Device: Alfapump

INTERVENTIONS:
Device: Alfapump — Implant Alfapump® System

SUMMARY:
1. Summary of Clinical Investigation

A summary of the clinical investigation is provided below and includes the primary objective of the study, the safety and feasibility endpoints, the number of subjects to be enrolled, the study duration, the subject follow-up and the inclusion/exclusion criteria.

1. Primary Objective

   The primary objective of the study is to evaluate the safety and feasibility of the alfapump® System indication for use in the management of fluid in NYHA Class III and ambulatory NYHA Class IV heart failure patients who have an eGFR of > 15 to < 60 mL/min/1.73m2.
2. Study Endpoints

   1. Primary Safety Endpoint

      The primary safety endpoint will be an assessment of the occurrence of adverse events (AEs) and serious adverse events (SAEs) related to:
      1. Surgical implant of the alfapump®
      2. Device malfunctions
      3. Dialysate infusion
   2. Secondary Safety Endpoints

      The secondary endpoint will be an assessment of:
      1. Time to first hospitalization related to fluid management after the activation of the alfapump® System and initiation of dialysate infusion has occurred
      2. Rate of occurrence of re-hospitalizations related to fluid management
      3. All-cause mortality
   3. Assessment of Feasibility for Fluid Management in Heart Failure Indication The feasibility of the alfapump® System for management of fluid in NYHA Class III and ambulatory NYHA Class IV heart failure patients with renal dysfunction will be assessed by the net fluid balance as measured by the ability of the alfapump® System to move more fluid to the bladder than dialysate instilled.

ELIGIBILITY:
Inclusion Criteria

* Males or females ≥ 18 years and < 80 years of age
* Patients exhibiting physical signs of excessive fluid retention (i.e. elevated JVD, peripheral edema, ascites, pulmonary edema, weight gain etc.)
* Patients with an eGFR by the Modification of Diet in Renal Disease (MDRD) of > 15 to < 60 mL/min/1.73m2
* Patients with a brain natriuretic peptide (BNP) ≥ 150 pg/mL and/or N-terminal prohormone of brain natriuretic peptide (NT-proBNP) ≥ 600 pg/mL at time of screening or BNP ≥ 100 pg/mL and/or NTproBNP ≥ 400 pg/mL
* Patients who have a Six Minute Walk Test (SMWT) exercise capacity between 100 and 400 meters
* Patients presenting with NYHA Class III or ambulatory NYHA Class IV heart failure who have been on optimal medical management (OMM) based on current heart failure practice guidelines and who are failing to respond to or cannot tolerate one or more of the following interventions:

  1. Treatment with diuretic therapy
  2. Treatment with angiotensin converting enzyme (ACE) inhibitors or angiotensin receptor blockers (ARBs) for at least 30 days
  3. Treatment with nitrates and/or vasodilators at the investigator's discretion
  4. Treatment with beta-blockers for at least 90 days
  5. Treatment with cardiac resynchronization therapy (CRT)
  6. Treatment with an automatic implantable cardioverter defibrillator (AICD)
* Patients who demonstrate compliance with the current medical regimen as reported by the treating physician

Enrollment Exclusion Criteria

* Patients presenting with acute decompensated heart failure requiring hospitalization for management of their symptoms (i.e. hospitalization for exacerbation of chronic heart failure manifested by signs and symptoms requiring intravenous and/or more aggressive therapy)
* Patients with ascites on physical examination resulting predominantly from right heart failure
* Patients who have an indication for and are candidates for CRT but who have not been treated with CRT
* Patients who have an indication for and are candidates for an AICD but who have not been implanted with an AICD
* Patients with reversible causes of heart failure which may be remedied by conventional surgery or other interventions
* Patients with an eGFR by MDRD < 15 or > 60 ml/min/1.73m2
* Patients with a body mass index (BMI) < 18 kg/m2or > 35 kg/m2
* Patients with severe pulmonary disease by history (i.e. severe chronic obstructive pulmonary disease, severe hypoxia or a pulmonary artery mean pressure >40 mm Hg)
* Patients who have experienced a myocardial infarction (MI) within the past 90 days
* Patients who have experienced a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 90 days
* Patients who have undergone cardiac surgery or other major surgery within the past 90 days
* Patients who are candidates for and require a concomitant surgical procedure [i.e. coronary artery bypass graft (CABG), valvular surgery, etc.
* Patients who are candidates for and require temporary or durable mechanical circulatory support [i.e. intra-aortic balloon pump (IABP), ventricular assist device (VAD), extracorporeal membrane oxygenation (ECMO)]
* Patients with confirmed untreated abdominal aortic aneurysm (AAA) > 5 cm in diameter diagnosed within the past six months
* Patients with active systemic or uncontrolled infections
* Patients who are pregnant (Note: Negative pregnancy test will be required in all women - Patients with known alcohol or illicit drug abuse or dependence within the previous three months
* Patients who are currently enrolled or who have participated in the past 30 days in another therapeutic and/or interventional clinical study
* Patients with technical obstacles that pose an inordinately high surgical risk in the judgment of the Investigator
* Patients who have any underlying condition that, in the opinion of the Investigator, would disqualify the patient for inclusion in the study, limit survival to less than one year, or not permit valid consideration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-31 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | Q1 2017 and Q3 2017
  4 weeks after the third patient implanted an initial safety review will be done and after the last patient completed 3 months of dialysate administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Military Hospital - State Health Centre, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided
Study cancelled, therefore not applicable at time of answering this remark.